CLINICAL TRIAL: NCT01989130
Title: Evaluation of the Cepheid Xpert CT/NG For Management of STI in the ED: Immediate V. Delayed Test Results
Brief Title: Evaluation of Immediate v. Delayed CT/NG Test for Treatment in the ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Cepheid (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 071346
Record Dates: First submitted 2013-11-06; First posted 2013-11-20 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Reproductive Tract Infections
Keywords: antimicrobial stewardship; Cepheid Xpert CT/NG; chlamydia; gonorrhea; emergency department; Diagnostic Techniques, Obstetrical and Gynecological; Diagnostic Techniques, Urological
MeSH Terms: conditions — Reproductive Tract Infections; Chlamydia Infections; Gonorrhea; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real-time results with Cepheid Xpert CT/NG Test (Experimental): Diagnosis of +/- CT/NG within 2 hours of specimen entering laboratory
  Interventions: Device: Cepheid Xpert CT/NG Test
- Batched results with Roche AMPLICOR CT/NG test (Active Comparator): Diagnosis of +/- CT/NG within 1 to 4 days of visit to the ED
  Interventions: Device: Roche AMPLICOR CT/NG

INTERVENTIONS:
Device: Roche AMPLICOR CT/NG
  Arms: Batched results with Roche AMPLICOR CT/NG test
Device: Cepheid Xpert CT/NG Test
  Arms: Real-time results with Cepheid Xpert CT/NG Test

SUMMARY:
The purpose of this study is to determine if immediate availability of GeneXpert® CT/NG test results reduces the overtreatment rate for ED patients with suspected gonorrhea or chlamydia and to assess changes in clinician management decisions with real-time test results.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial in patients aged 18 and older where the treating clinician is ordering a CT/NG test. Clinicians will be approached by a research assistant while they are in the ED and asked whether a CT/NG swab will be ordered and if CT/NG is in the differential diagnosis. Then, potentially eligible patients will be approached and asked for consent to enroll. For patients that consent, simple randomization procedure (i.e. random number generator) will be used to assign patients to either immediate test results or delayed test results. Typically, in the ED these tests are ordered for diagnostic rather than screening purposes (symptoms of vaginal discharge, abdominal pain, etc). Patients will be randomized to batched testing with the Roche AMPLICOR CT/NG (standard of care, control group) or immediate testing of clinical specimens with Cepheid CT/NG with real-time result reporting (within 90 minutes) to the treating clinician in the ED. Patient interview and clinician survey will be conducted to ascertain perceptions of illness and the test. A follow up interview will be conducted with the patient to determine clinical and public health outcomes.

A validation of the Cepheid CT/NG test will be conducted against the hospital standard of care on </= 40 pilot participants. Pilot participants will be asked to provide 2 endocervical swabs and a urine specimen. All surveys and interviews will be conducted on pilot patients.

While many outcomes can be measured in this study, the investigators will power this study to reduce the overtreatment rate with antibiotics. Assuming a baseline overtreatment rate of 88% (# treated with antibiotics/# without disease), to reduce this rate by 50% (to 44%), at a power of 80% and alpha of 0.05, the investigators will need to enroll 42 patients (21 controls and 21 study patients) with negative tests. Given an estimated positive rate of 6%, and that approximately 50% of patients who receive these tests for any reason will be treated empirically with antibiotics, the investigators think that enrolling a total of 70 patients with full data (enrollment survey, clinician survey, and follow up survey) would be sufficient to identify trends with this subject matter. Due to the sensitive nature of the subject matter and the high percentages of lost-to-follow up with ED patients, the investigators estimate approximately 50% will have incomplete data. Therefore, the investigators request to enroll 150 patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years
* clinical suspicion of CT/NG
* able to give informed consent
* willingness to wait for test result

Exclusion Criteria:

* less than 18 years
* pregnancy
* prisoners
* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa May, MD, Principal Investigator — George Washington University
Locations (1):
- The George Washington University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Andric B, Drowos J, Trepka MJ, Suciu G, Alonso A, Hennekens CH. High frequencies of negative pretreatment results following presumptive antibiotic treatment for chlamydia and gonorrhea. South Med J. 2013 May;106(5):321-6. doi: 10.1097/SMJ.0b013e318291b3c2. PMID 23644641
- [Background] Levitt MA, Johnson S, Engelstad L, Montana R, Stewart S. Clinical management of chlamydia and gonorrhea infection in a county teaching emergency department--concerns in overtreatment, undertreatment, and follow-up treatment success. J Emerg Med. 2003 Jul;25(1):7-11. doi: 10.1016/s0736-4679(03)00131-8. PMID 12865101
- [Background] Gaydos CA, Van Der Pol B, Jett-Goheen M, Barnes M, Quinn N, Clark C, Daniel GE, Dixon PB, Hook EW 3rd; CT/NG Study Group. Performance of the Cepheid CT/NG Xpert Rapid PCR Test for Detection of Chlamydia trachomatis and Neisseria gonorrhoeae. J Clin Microbiol. 2013 Jun;51(6):1666-72. doi: 10.1128/JCM.03461-12. Epub 2013 Mar 6. PMID 23467600
- [Derived] May L, Ware CE, Jordan JA, Zocchi M, Zatorski C, Ajabnoor Y, Pines JM. A Randomized Controlled Trial Comparing the Treatment of Patients Tested for Chlamydia and Gonorrhea After a Rapid Polymerase Chain Reaction Test Versus Standard of Care Testing. Sex Transm Dis. 2016 May;43(5):290-5. doi: 10.1097/OLQ.0000000000000438. PMID 27100764

RESULTS

PARTICIPANT FLOW:
Groups:
- Real-time Results With Cepheid Xpert CT/NG Test: Diagnosis of +/- CT/NG within 2 hours of specimen entering laboratory
  Cepheid Xpert CT/NG Test
- Batched Results With Roche AMPLICOR CT/NG Test: Diagnosis of +/- CT/NG within 1 to 4 days of visit to the ED
  Roche AMPLICOR CT/NG
Period: Overall Study
Arm/Group | Real-time Results With Cepheid Xpert CT/NG Test | Batched Results With Roche AMPLICOR CT/NG Test
Started | 43 | 27
Completed | 43 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real-time Results With Cepheid Xpert CT/NG Test | Batched Results With Roche AMPLICOR CT/NG Test | Total
Number analyzed (Participants) | 43 | 27 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 41 | 26 | 67
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 16 | 43
  Male | 16 | 11 | 27
Region of Enrollment [Number; unit: participants]
  United States | 43 | 27 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Prescribed Antibiotic Treatment
Description: Measurement of the number and type of antibiotics prescribed to CT/NG + v. CT/NG - in both groups
Time Frame: one year
Measure: Number; unit: percentage of 70 participants
Arm/Group | Real-time Results With Cepheid Xpert CT/NG Test | Batched Results With Roche AMPLICOR CT/NG Test
Number analyzed (Participants) | 43 | 27
percentage of 70 participants | 7.1 | 5.7

2. Primary Outcome: Health Utilization
Description: Number of participants with visits to healthcare facilities/providers and non-ED related medications purchased in 7-10 days after enrollment
Time Frame: one year
Population: Analysis included patients that responded to the 7-10 day follow-up phone call.
Measure: Count of Participants; unit: Participants
Arm/Group | Real-time Results With Cepheid Xpert CT/NG Test | Batched Results With Roche AMPLICOR CT/NG Test
Number analyzed (Participants) | 20 | 17
Participants
  Subsequent hospitalization | 1 | 1
  subsequent office visit | 5 | 2
  new prescription drugs | 3 | 0

3. Primary Outcome: Healthcare Cost
Description: To quantify the amount billed to insurance companies and out of pocket expenses for initial encounter
Time Frame: one year
Population: This outcome measure was not measured, as insurance coverage for hospital and physician charges was unavailable.
Arm/Group | Real-time Results With Cepheid Xpert CT/NG Test | Batched Results With Roche AMPLICOR CT/NG Test
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Resolution of Symptoms
Description: Number of patients that report having no symptoms 7 to 10 days after initial encounter
Time Frame: one year
Population: Analysis of patients who completed the 7-10 day follow-up phone call
Measure: Count of Participants; unit: Participants
Arm/Group | Real-time Results With Cepheid Xpert CT/NG Test | Batched Results With Roche AMPLICOR CT/NG Test
Number analyzed (Participants) | 20 | 17
Participants | 17 | 10

ADVERSE EVENTS:
Arm/Group | Real-time Results With Cepheid Xpert CT/NG Test | Batched Results With Roche AMPLICOR CT/NG Test
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No